CLINICAL TRIAL: NCT05208554
Title: Feasibility and Acceptability of a Dyad-based Physical Activity Intervention for Hematopoietic Cell Transplant Recipients and Caregivers
Brief Title: Physical Activity Intervention for Hematopoietic Cell Transplant Recipients and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Nandita Khera, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-007867; NCI-2022-02761 (Registry Identifier: NCI)
Record Dates: First submitted 2022-01-04; First posted 2022-01-26 (Actual); Last update posted 2025-05-19 (Actual); Status verified 2025-05

CONDITIONS: Hematopoietic Cell Transplant
Keywords: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Family-Focused Facilitated Fitness program (Experimental): Couple-based physical activity intervention commencing 14 (+/-7) days post-transplant (8 sessions with a health counselor). Sessions 1-4 will train couples in the use of communal coping strategies to support one another in achieving PA goals. Skill building will focus on instruction and practice in adaptive communication, with emphases on adaptive speaking, responsive listening, and joint decision-making and problem-solving around PA. Instruction and practice will focus specifically on communication about PA and working together (we versus me) to increase PA. Sessions 5-8 will afford check-in, review of PA progress, and troubleshooting any barriers to PA. All sessions will be dyad-based but will include delivery of individualized step goals for the next week using an adaptive approach and based on remotely-monitored Fitbit step data. Specifically, the 75th percentile rank of each participant's last 7 days of recorded days will serve as the step goal prescription for the next week.
  Interventions: Behavioral: Integrated health counseling and step prescription

INTERVENTIONS:
Behavioral: Integrated health counseling and step prescription — 8 weekly dyad-based sessions with a health counselor to train couples in the use of communal coping strategies to support one another in achieving physical activity goals plus individualized step prescription based on remotely-monitored Fitbit-derived step counts the week prior

SUMMARY:
Levels of physical activity (PA) among cancer survivors are low, yet PA may ameliorate effects of treatment (Phillips et al., 2014). We focus here on PA following the most intensive form of cancer treatment, hematopoietic cell transplantation (HCT), with multiple sequelae including graft-versus-host disease and cardiovascular and pulmonary complications. PA is diminished post-transplant (Hacker & Mjukian, 2014; Morishita et al., 2017). This decrease is associated with poorer physical functioning (Bennett et al., 2016), in turn associated with greater mortality (Wood et al., 2016). Moderate exercise has been deemed safe for HCT patients (Wiskemann et al., 2014), and PA interventions feasible (Hacker & Mjukian, 2014). Findings regarding efficacy are mixed, largely due to heterogeneity of intervention components and outcomes (Liu et al., 2009; Persoon et al., 2013). All PA interventions in the HCT setting have focused entirely on patients, ignoring an opportunity to synergistically engage and benefit the caregiver, a 24/7 role requiring provision of medical, logistical, and emotional support. Distress is common among HCT caregivers and their own health promotion is neglected (Applebaum et al., 2016). In addition, the patient-caregiver relationship can be compromised, and communication patterns disrupted (Langer et al., 2009). Guided by interdependence (Kelley et al., 1983) and communal coping (Lyons et al., 1998) perspectives, our 8-session PA intervention provides training in communication skills and behavior change techniques to help patient-caregiver dyads support one another in PA. Previous testing with a sample of breast cancer and prostate cancer survivors and caregivers demonstrated feasibility, but relied solely on self-reported PA and self-determined PA goals (Porter et al., 2018). We have adapted this protocol for HCT and will use a wearable device, a Fitbit tracker, to objectively monitor PA and to provide participants with weekly individualized step goals.

Specific aims are to: (1) determine feasibility of adherence to a dyad-based PA intervention (# of sessions attended and Fitbit wear adherence) for HCT recipients and caregivers (15 dyads) using a single-group pre-post design; (2) determine acceptability of the intervention (dimensions of treatment satisfaction); and (3) describe patterns of change in PA and communal coping from baseline to follow-up. Findings will inform the design of a randomized controlled trial to test efficacy of the intervention to improve physical endurance and relational well-being.

ELIGIBILITY:
Inclusion Criteria - Patients:

* Scheduled to receive an autologous or allogeneic HCT.
* Being married or in a committed cohabiting relationship.
* English speaking and comprehending.
* Physician approval to participate in a walking program.

Inclusion Criteria - Caregivers:

* Married to or in a cohabiting relationship with the patient.
* Able to participate in a walking program.

Exclusion Criteria - Patients:

* Not scheduled to receive an HCT or already post-HCT.
* Unmarried or not in a committed cohabiting relationship.
* Non-English speaking and comprehending.
* Not medically approved to participate in walking program.
* Enrolled in competing behavioral intervention.

Exclusion Criteria - Caregivers:

* Not married to or partnered/ cohabiting with the patient.
* Unable to participate in a walking program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Treatment adherence | 8 weeks
  Percentage of couples attending all 8 intervention sessions
Fitbit adherence | 7 days
  Percentage of participants providing valid wear data 4 of 7 days/ week during assessment periods (device worn >=10 hours/ day)

SECONDARY OUTCOMES:
Treatment satisfaction | 90-100 days post-transplant
  Multi-Dimensional Treatment Satisfaction Measure

CONTACTS AND LOCATIONS:
Overall Officials: Nandita Khera, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Pheonix, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials